CLINICAL TRIAL: NCT02640248
Title: Endotracheal Tube Intracuff Pressure and Leak Around the Cuff During Retractor Placement for Adenotonsillectomy
Status: Withdrawn | Type: Observational
Why Stopped: Original PI left NCH, study never started then
Sponsor: Kris Jatana (Other)
Responsible Party: Sponsor-Investigator, Kris Jatana, Ears Nose Throat Surgeon, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00902
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2019-11

CONDITIONS: Otolaryngological Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cuff ETT
  Interventions: Device: Cuff ETT

INTERVENTIONS:
Device: Cuff ETT

SUMMARY:
The investigators have devised a simple method to continuously measure the CP using an invasive pressure monitoring setup (IPMS), which is used routinely in the operating room to monitor arterial or central venous pressures. The investigators have previously confirmed both in vitro and in vivo (previous IRB approved protocol), a clinically applicable agreement of the IPMS readings with the values obtained from a standard manometer (gold standard). In the current study, we will prospectively evaluate the relationship between the patient's head position and CP in patients undergoing otolaryngological surgery and also measure the oxygen concentration in the oropharynx to determine the potential risk of an airway fire.

ELIGIBILITY:
Inclusion Criteria:

* Less than 18 years of age, undergoing otolaryngological surgery with endotracheal intubation

Exclusion Criteria:

* Patient who is intubated with an uncuffed endotracheal tube
* Patients who have a limitation for movement of the neck or concerns of the stability of the cervical spine.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Less than 18 years of age, undergoing otolaryngological surgery with endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Changes in intracuff pressure | during time of surgery
  Changes in intracuff pressure of cuffed ETT related to the position of the patient's head and retractor placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States